CLINICAL TRIAL: NCT03133104
Title: Retrospective Review of Repeat Antenatal Corticosteroids in Preterm Premature Rupture of Membranes
Brief Title: Repeat Antenatal Corticosteroids
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Cara Buskmiller, MD, Principal Investigator, St. Louis University
Other Study IDs: 27833
Record Dates: First submitted 2017-01-17; First posted 2017-04-28 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Antenatal Corticosteroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- antenatal corticosteroids: Women who received a rescue dose of steroids
  Interventions: Other: Antenatal corticosteroids
- No antenatal corticosteroids: Women who did not received a rescue dose of steroids

INTERVENTIONS:
Other: Antenatal corticosteroids — Women and neonates with PPROM who received a repeat dose of antenatal corticosteroids, compared to women with PPROM who did not received a repeat course of antenatal corticosteriods
  Groups: antenatal corticosteroids

SUMMARY:
This study will review records of women who broke their water early who received a repeat course of antenatal steroids.

DETAILED DESCRIPTION:
Antenatal corticosteroids (ANCS) administered to a mother at risk of preterm delivery have been shown to decrease morbidity of prematurity if preterm birth occurs. Although early animal studies found that many repeated doses led to growth restriction a single repeat dose was found to benefit human neonates without a significant decrease in birth weight.

Current guidelines recommend two doses of ANCS administered 24 hours apart as a single "course." A repeat course of steroids is administered no less than 1-2 weeks after the first course if the mother remains at risk of preterm delivery. However, the main studies supporting the repeat course of ANCS excluded women with preterm premature rupture of membranes (PPROM). These authors designed exclusion criteria this way because of a theoretical increased risk of chorioamnionitis with administration of a glucocorticoid, which may have immunosuppressant effects. As a result, there is insufficient data to recommend a repeat dose of ANCS in women with PPROM.

One study and its follow up publication did include women with PPROM. It did not find an increased incidence of chorioamnionitis between the treatment and the placebo groups, although women with PPROM were not analyzed separately.

The combination of no increased incidence of chorioamnionitis but no clearly studied populations creates an opportunity for a randomized controlled trial of repeat doses of ANCS including only women with PPROM.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preterm premature rupture of membranes

Exclusion Criteria:

* Women who did not have preterm premature rupture of membranes

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pregnant women preterm premature rupture of membranes All ethnic backgrounds
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2017-01-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Infant outcomes | 1 year
  infant birth weight

CONTACTS AND LOCATIONS:
Overall Officials: Cara Buskmiller, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No